CLINICAL TRIAL: NCT05375929
Title: A RANDOMIZED, OPEN-LABEL, PARALLEL-GROUP STUDY TO EVALUATE THE SAFETY AND EFFICACY OF ABROCITINIB 100 MG AND 200 MG TABLETS IN PARTICIPANTS AGED 12 YEARS AND OLDER WITH MODERATE TO SEVERE ATOPIC DERMATITIS IN INDIA
Brief Title: A Study to Learn About Abrocitinib Tablets in People With Atopic Dermatitis in India
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B7451094
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Atopic Dermatitis
Keywords: AD; Atopic Eczema
MeSH Terms: conditions — Dermatitis, Atopic | interventions — abrocitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abrocitinib 100 mg (Experimental): Participants will receive abrocitinib 100 mg by mouth (QD).
  Interventions: Drug: Abrocitinib 100 mg
- Abrocitinib 200 mg (Experimental): Participants will receive abrocitinib 200 mg QD.
  Interventions: Drug: Abrocitinib 200 mg

INTERVENTIONS:
Drug: Abrocitinib 100 mg — Orally administered, abrocitinib 100 mg tablets QD
  Arms: Abrocitinib 100 mg
Drug: Abrocitinib 200 mg — Orally administered, abrocitinib 200 mg tablets QD.
  Arms: Abrocitinib 200 mg

SUMMARY:
The purpose of this clinical trial is to learn about the safety and how well the study medicine (called Abrocitinib) works for the potential treatment of moderate to severe Atopic Dermatitis (AD) in India. AD, also known as atopic eczema, is a chronic, relapsing skin condition characterized by dry, itchy skin lesions which can affect any part of the body. Adult peoples who participate in this study will take either 100 mg or 200 mg of abrocitinib tablets by mouth for a duration of 12 weeks and adolescents will take for duration of 52 weeks. Knee Magnetic Resonance Imagine (MRI) will be done on adolescent peoples to determine bone safety findings. We will examine the experiences of people receiving the study medicines. This will help us determine if the study medicines are safe and how well they work.

DETAILED DESCRIPTION:
Abrocitinib is an oral, once daily Janus kinase 1 (JAK1) selective inhibitor for the treatment of moderate to severe Atopic Dermatitis (AD). Selective inhibition of JAK1 with abrocitinib modulates signaling by Interleukin-4 (IL-4), Interleukin (IL-13), and other cytokines [eg, IL-31, IL-22, and thymic stromal lymphopoietin (TSLP)] involved in the pathogenesis of Atopic Dermatitis and pruritus.

This is a randomized, open label, parallel group study to assess the safety and efficacy of orally administered tablets of abrocitinib in participants aged 12 years and older with moderate to severe AD in India. There is a planned treatment duration of 12 weeks, with 4 weeks of off-treatment safety follow up thereafter.

This study protocol also includes a sub-study evaluating whether abrocitinib has any potential effects on adolescent bone with regard to abnormal bone findings in knee magnetic resonance imaging (MRI). Adolescent participants (12 to <18 years of age) will continue to receive study intervention until 1 year after randomization into the main study.

ELIGIBILITY:
Inclusion Criteria:

This study is seeking participants who:

1. Must be of 12 years of age or older, at the time of informed consent.
2. Meet all the following Atopic Dermatitis (AD) criteria:

   * Clinical diagnosis of chronic AD (also known as atopic eczema) for at least 1 year prior to Day 1 and has confirmed AD (Hanifin and Rajka criteria of AD10).
   * Moderate to severe AD (affected body surface area (BSA) ≥10%, Investigator's Global Assessment (IGA) ≥3, Eczema Area and Severity Index (EASI) ≥16, and Peak Pruritus Numerical Rating Scale (PP-NRS) ≥4 at the baseline visit);
   * Documented recent history (within 6 months before the screening visit) of inadequate response to treatment with topical medications for at least 4 weeks, or for whom topical treatments are otherwise medically inadvisable (eg, because of important side effects or safety risks), or who have required systemic therapies for control of their disease.
3. Negative pregnancy test for females of childbearing potential at Screening. Female participants of childbearing potential must agree to use a highly effective method of contraception for the duration of the active treatment period and for at least 28 days after the last dose of study intervention.
4. Body weight ≥25 kg at Baseline
5. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the Informed Consent Document (ICD) and in this protocol. Evidence of a personally signed and dated ICD indicating that the participant (or a legally acceptable representative, parent(s)/legal guardian) has been informed of all pertinent aspects of the study. For minors under the age of legal consent in India, assent of the participating child needs to be documented for the age range 12 to 18 years in addition to the parental informed consent.

Exclusion Criteria:

This study does not include participants who:

1. Currently have active forms of other inflammatory skin diseases or have evidence of skin conditions (eg, psoriasis, seborrheic dermatitis, lupus).
2. A current or past medical history of conditions associated with thrombocytopenia, coagulopathy or platelet dysfunction or QT interval abnormalities.
3. Have increased risk of developing venous thromboembolism, eg, deep vein thrombosis or pulmonary embolism:
4. Have a history of any lymphoproliferative disorder such as Epstein Barr virus (EBV) related lymphoproliferative disorder, history of lymphoma, leukemia, or signs or symptoms suggestive of current lymphatic or lymphoid disease.
5. Past history or active infection with Mycobacterium tuberculosis (TB), disseminated herpes zoster or disseminated herpes simplex, human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C.
6. Have any malignancies or have a history of malignancies with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ.
7. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgement, make the participant inappropriate for the study. Any psychiatric condition including recent or active suicidal ideation or behavior that met any of the following criteria when screened for during the main study:

   * Suicidal ideation associated with actual intent and a method or plan in the past year: "Yes" answers on items 4 or 5 of the Columbia suicide severity rating scale (C-SSRS);
   * Previous history of suicidal behaviors in the past 5 years: "Yes" answer (for events that occurred in the past 5 years) to any of the suicidal behavior items of the C-SSRS;
   * Any lifetime history of serious or recurrent suicidal behavior;
   * The presence of any current major psychiatric disorder that is not explicitly permitted in the inclusion/exclusion criteria;
   * In the opinion of the investigator or Pfizer (or designee) exclusion is required.
8. Prior treatment with systemic janus kinase (JAK) inhibitors.
9. Participants who are vaccinated with live attenuated vaccine within the 6 weeks prior to the first dose of abrocitinib or who are expected to be vaccinated with these vaccines during treatment or during the 6 weeks following discontinuation of abrocitinib.
10. Have received any of the following treatment regimens specified in the timeframes outlined below:

    Within 1 year of first dose of study intervention:
    * Prior treatment with non B cell-specific lymphocyte depleting agents/therapies (eg, alkylating agents [eg, cyclophosphamide or chlorambucil], total lymphoid irradiation, etc.). Participants who have received rituximab or other selective B lymphocyte depleting agents (including experimental agents) are eligible if they have not received such therapy for at least 1 year prior to study baseline and have normal cluster of differentiation (CD) 19/20+ counts by fluorescence activated cell sorting (FACS) analysis.

    Within 12 weeks of first dose of study intervention:
    * Biologic drugs that have immunomodulatory properties or could be used to treat AD: within 12 weeks of first dose of investigational product or 5 half-lives (if known), whichever is longer.

    Other biologics without immunomodulatory properties (eg, insulin) are permissible at the judgement of the Investigator.

    Within 4 weeks of first dose of study intervention:
    * Use of oral immunosuppressive drugs (eg, Cyclosporine A (CsA), azathioprine, methotrexate, systemic corticosteroids, mycophenolate mofetil, Interferon gamma) within 4 weeks of first dose of study intervention or within 5 half-lives (if known), whichever is longer.

    NOTE: Systemic corticosteroids must be discontinued before Study Day 1, but a specific timeframe for discontinuation prior to first dose of abrocitinib is not required.

    NOTE: Corticosteroid inhalers and intranasal sprays are permissible. NOTE: Ophthalmic corticosteroids are permissible.

    Within 1 week of first dose of study intervention:
    * Anti-platelet drugs. Note: low dose acetyl salicylic acid (<100 mg once daily [QD]) is permitted, for the purpose of cardiovascular prophylaxis, at the discretion of the investigator.
11. Require treatment with prohibited concomitant medication(s) or have received a prohibited concomitant medication.
12. Participation in other studies involving investigational drug(s) or vaccine within 8 weeks or within 5 half-lives (if known) whichever is longer, prior to study entry and/or during study participation.
13. Any of the following abnormalities in clinical laboratory tests at Screening:

    * Absolute neutrophil count of <1.0 × 109/L (<1000/mm3);
    * Platelet count of <150 × 109/L (<150,000/mm3);
    * Absolute lymphocyte count of <0.50 × 109/L (<500/mm3);
    * Estimated Creatinine Clearance <60 mL/min using the Cockcroft Gault method;
    * Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) values >2 times the Upper Limit of Normal (ULN);
    * Total Bilirubin (TBili) ≥1.5 times the ULN.
14. Pregnant or breastfeeding women, or women of childbearing potential who are unwilling to use highly effective contraception consistently and correctly for the entire duration of the study and for at least 28 days after the last dose of study intervention.
15. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-07-16 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2024-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- India (15):
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - Government Medical College & Shri Sayajirao General Hospital, Vadodara, Gujarat
  - RajaRajeswari Medical College and Hospital, Bengaluru, Karnataka
  - Father Muller Medical College Hospital, Mangalore, Karnataka
  - Mahatma Gandhi Mission's Medical College & Hospital, Aurangabad, Maharashtra
  - Orange City Hospital and Research Institute, Nagpur, Maharashtra
  - Assured Care Plus Hospital, Nashik, Maharashtra
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - S. P. Medical College & A. G. Hospitals, Bikaner, Rajasthan
  - Apex Hospitals Pvt. Ltd., Jaipur, Rajasthan
  - Calcutta School of Tropical Medicine, Kolkata, West Bengal
  - Postgraduate Institute of Medical Education & Research, Chandigarh
  - Maharaja Agrasen Hospital, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 200 participants aged greater than or equal to (>=) 12 years with moderate to severe atopic dermatitis (AD) were enrolled in the study.
Pre-assignment Details: This study had main study and substudy. Adolescent participants consented for substudy at main study inform consent/assent. Eligible participants who consented for substudy continued to receive study intervention as assigned in the main study after the 12-week treatment period, until 1 year after randomization in the main study or until they turned 18 years of age. As per statistical analysis plan (SAP) participants' disposition, and discontinuation were to be summarized by treatment arm.
Groups:
- Main Study: Abrocitinib 200 mg QD: Participants received abrocitinib 200 milligram (mg), orally once daily (QD) for 12 weeks.
- Main Study: Abrocitinib 100 mg QD: Participants received abrocitinib 100 mg, orally QD for 12 weeks.
- Substudy: Abrocitinib 200 mg: Eligible adolescent participants who received abrocitinib 200 mg orally QD for 12 weeks in main study and continued to receive the same treatment in similar way until 1 year after randomization (on Day 1) from main study.
- Substudy: Abrocitinib 100 mg: Eligible adolescent participants who received abrocitinib 100 mg orally QD for 12 weeks in main study and continued to receive the same treatment in similar way until 1 year after randomization (on Day 1) from main study.
Period: Main Study: Treatment Phase (12 Weeks)
Arm/Group | Main Study: Abrocitinib 200 mg QD | Main Study: Abrocitinib 100 mg QD | Substudy: Abrocitinib 200 mg | Substudy: Abrocitinib 100 mg
Started | 99 | 101 (1 participant was randomized to 200 mg arm but received 100 mg, hence included here.) | 0 | 0
Safety Analysis Set (According to actual treatment that participants received.) | 99 (Participants received 200 mg QD.) | 101 (Participants received 100 mg QD.) | 0 | 0
Full Analysis Set (According to the treatment arm participants were randomized to.) | 100 (Participants randomized to 200 mg QD arm.) | 100 (Participants randomized to 100 mg QD arm.) | 0 | 0
Completed | 91 | 94 | 0 | 0
Not Completed | 8 | 7 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 5 | 0 | 0
Not completed — Withdrawal by parent/guardian | 0 | 1 | 0 | 0
Period: Main Study: Follow-up (4 Weeks)
Arm/Group | Main Study: Abrocitinib 200 mg QD | Main Study: Abrocitinib 100 mg QD | Substudy: Abrocitinib 200 mg | Substudy: Abrocitinib 100 mg
Started | 91 | 94 | 0 | 0
Completed | 90 | 93 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Did not complete study follow-up | 0 | 1 | 0 | 0
Period: Substudy: Treatment Phase (1 Year)
Arm/Group | Main Study: Abrocitinib 200 mg QD | Main Study: Abrocitinib 100 mg QD | Substudy: Abrocitinib 200 mg | Substudy: Abrocitinib 100 mg
Started | 0 (Period is for substudy.) | 0 (Period is for substudy.) | 19 (Only eligible adolescents participants who consented continued treatment in substudy.) | 16 (Only eligible adolescents participants who consented continued treatment in substudy.)
Completed | 0 | 0 | 12 | 15
Not Completed | 0 | 0 | 7 | 1
Not completed — Withdrawal by parent/guardian | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0
Period: Substudy: Follow-up (4 Weeks)
Arm/Group | Main Study: Abrocitinib 200 mg QD | Main Study: Abrocitinib 100 mg QD | Substudy: Abrocitinib 200 mg | Substudy: Abrocitinib 100 mg
Started | 0 | 0 | 17 (Participants who were followed-up.) | 15
Completed | 0 | 0 | 17 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention and who had taken at least 1 dose of study intervention. Participants were analyzed according to the treatment they actually received. Substudy analysis set (SAS) included all participants who entered the substudy and who took at least 1 dose of study intervention during the substudy.
Groups:
- Main Study: Abrocitinib 200 mg QD: Participants received at least 1 dose of abrocitinib 200 mg, orally QD in the study.
- Main Study: Abrocitinib 100 mg QD: Participants received at least 1 dose of abrocitinib 100 mg, orally QD in the study.
- Total: Total of all reporting groups
Arm/Group | Main Study: Abrocitinib 200 mg QD | Main Study: Abrocitinib 100 mg QD | Total
Number analyzed (Participants) | 99 | 101 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The number analyzed in sub study refers to the number of participants enrolled in sub study.
  Years
    Main Study | 35.37 (17.19) | 37.50 (17.49) | 36.45 (17.33)
    Substudy: number analyzed (Participants) | 19 | 16 | 35
    Substudy | 14.79 (2.25) | 14.44 (1.36) | 14.63 (1.88)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed in sub study refers to the number of participants enrolled in sub study.
  Participants
    Main Study: Female | 61 | 48 | 109
    Main Study: Male | 38 | 53 | 91
    Substudy: number analyzed (Participants) | 19 | 16 | 35
    Substudy: Female | 12 | 7 | 19
    Substudy: Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed in sub study refers to the number of participants enrolled in sub study.
  Participants
    Main Study: Hispanic or Latino | 0 | 0 | 0
    Main Study: Not Hispanic or Latino | 99 | 101 | 200
    Main Study: Unknown or Not Reported | 0 | 0 | 0
    Substudy: number analyzed (Participants) | 19 | 16 | 35
    Substudy: Hispanic or Latino | 0 | 0 | 0
    Substudy: Not Hispanic or Latino | 19 | 16 | 35
    Substudy: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed in sub study refers to the number of participants enrolled in sub study.
  Participants
    Main Study: American Indian or Alaska Native | 0 | 0 | 0
    Main Study: Asian | 99 | 101 | 200
    Main Study: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Main Study: Black or African American | 0 | 0 | 0
    Main Study: White | 0 | 0 | 0
    Main Study: More than one race | 0 | 0 | 0
    Main Study: Unknown or Not Reported | 0 | 0 | 0
    Substudy: number analyzed (Participants) | 19 | 16 | 35
    Substudy: American Indian or Alaska Native | 0 | 0 | 0
    Substudy: Asian | 19 | 16 | 35
    Substudy: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Substudy: Black or African American | 0 | 0 | 0
    Substudy: White | 0 | 0 | 0
    Substudy: More than one race | 0 | 0 | 0
    Substudy: Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs): Main Study
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic or other situations where medical or scientific judgement should be exercised by investigator. AEs included SAEs and all non-SAEs.
Time Frame: From Day 1 of dosing up to 4 weeks post last dose (maximum up to Week 16)
Population: Safety analysis set included all participants randomly assigned to study intervention and who had taken at least 1 dose of study intervention. Participants were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Main Study: Abrocitinib 200 mg: Participants received abrocitinib 200 mg, orally QD for 12 weeks.
- Main Study: Abrocitinib 100 mg: Participants received abrocitinib 100 mg, orally QD for 12 weeks.
Arm/Group | Main Study: Abrocitinib 200 mg | Main Study: Abrocitinib 100 mg
Number analyzed (Participants) | 99 | 101
Participants
  AEs | 30 | 26
  SAEs | 0 | 1

2. Secondary Outcome: Percentage of Participants Who Achieved Investigator's Global Assessment (IGA) Score of Clear (0) or Almost Clear (1) and >= 2 Points Improvement From Baseline at Week 12: Main Study
Description: IGA assesses severity of AD on a 5-point scale (0 to 4: higher scores = more severity). Scores: 0= clear (no AD inflammatory signs except for any residual discolouration [post-inflammatory hyperpigmentation and/or hypopigmentation]); 1= almost clear (AD not entirely cleared- light pink residual lesions [except post-inflammatory hyperpigmentation], just barely perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting); 2= mild (AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting); 3= moderate (AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting); 4= severe (AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting). >=2 points improvement from baseline: decrease of at least 2 points in IGA score from baseline at Week 12.
Time Frame: Baseline (prior to dosing on Day 1), Week 12
Population: Full analysis set (FAS) included all participants randomly assigned to study intervention and who had taken at least 1 dose of study intervention. Participants were analyzed according to the treatment arm they were randomized to. Non-responder imputation (NRI) was applied. "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: Abrocitinib 200 mg | Main Study: Abrocitinib 100 mg
Number analyzed (Participants) | 99 | 100
Percentage of participants | 48.5 [38.6 to 58.3] | 50.0 [40.2 to 59.8]

3. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index (EASI) Response >= 75% Improvement From Baseline at Week 12: Main Study
Description: EASI evaluates severity of participant's AD based on both severity of lesion clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema [E], induration/papulation [I], excoriation [Ex] and lichenification [L]) scored separately for each of 4 body regions (head and neck [h], upper limbs [u], trunk [t]-[including axillae and groin] and lower limbs [l]-[including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh + Ih + Exh + Lh) + 0.2*Au*(Eu + Iu + ExU + Lu) + 0.3*At*(Et + It + Ext + Lt) + 0.4*Al*(El + Il + Exl +Ll); A = EASI area score. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD. >=75% improvement from baseline: decrease of 75% in EASI score from Baseline at Week 12.
Time Frame: Baseline (prior to dosing on Day 1), Week 12
Population: FAS included all participants randomly assigned to study intervention and who had taken at least 1 dose of study intervention. Participants were analyzed according to the treatment arm they were randomized to. NRI was applied. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: Abrocitinib 200 mg | Main Study: Abrocitinib 100 mg
Number analyzed (Participants) | 99 | 100
Percentage of participants | 71.7 [62.8 to 80.6] | 69.0 [59.9 to 78.1]

4. Secondary Outcome: Percentage of Participants Achieving Scoring Atopic Dermatitis (SCORAD) Response >= 75% Improvement From Baseline at Week 12: Main Study
Description: SCORAD: scoring index for AD combining extent (A), severity (B), subjective symptoms (C). A: rule of 9 was used to calculate BSA affected by AD as a % of whole BSA for each body region- head and neck 9%; upper limbs 9% each; lower limbs 18% each; anterior trunk 18%; back 18%; 1% for genitals. Score for each body region was added to determine A (0-100). B: severity of each sign (erythema; edema; oozing; excoriation; lichenification; dryness) assessed as none =0, mild =1, moderate =2, severe =3. Severity scores were added to give B (0-18). C: pruritus and sleep, each was scored by participant/caregiver using visual analogue scale (VAS) where 0= no itch/no sleeplessness and 10= worst imaginable itch/sleeplessness. Scores for itch and sleeplessness were added to give C (0-20). Total SCORAD was calculated: A/5 + 7*B/2 + C; total SCORAD range from 0-103; higher SCORAD scores = greater severity of AD. >=75% improvement from baseline: decrease of 75% in SCORAD score from Baseline at Week 12.
Time Frame: Baseline (prior to dosing on Day 1), Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: Abrocitinib 200 mg | Main Study: Abrocitinib 100 mg
Number analyzed (Participants) | 99 | 100
Percentage of participants | 47.5 [37.6 to 57.3] | 43.0 [33.3 to 52.7]

5. Secondary Outcome: Change From Baseline in Patient-Oriented Eczema Measure (POEM) Score at Weeks 2, 4, 8 and 12: Main Study
Description: POEM is a 7-item participant reported outcome (PRO) measure to assess the impact of AD over the past week. Items were: dryness or roughness of skin in day, skin being itchy in day, skin flaking off in day, skin cracking in day, skin bleeding in day, skin weeping or oozing in day and sleep disturbed in night. Each item is scored from 0 to 4, depending on number of days/night (for sleep items) over the past week symptoms happened, where 0= no days, 1= "1-2 days", 2= "3-4 days", 3= "5-6 days" and 4= "every day". Scores from all items are added up, which results in POEM score, ranging from 0 to 28, where higher scores indicate greater severity of AD and greater symptom burden.
Time Frame: Baseline (prior to dosing on Day 1), Weeks 2, 4, 8 and 12
Population: FAS evaluated. Participants were analyzed according to the treatment arm they were randomized to. All participants reported under "Number of Participants Analyzed" contributed data to the table but may not have evaluable data for every row. "Number Analyzed" signifies number of participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Main Study: Abrocitinib 200 mg | Main Study: Abrocitinib 100 mg
Number analyzed (Participants) | 100 | 100
Units on a scale
  Week 2: number analyzed (Participants) | 97 | 98
  Week 2 | -6.3 (4.97) | -5.1 (5.12)
  Week 4: number analyzed (Participants) | 96 | 96
  Week 4 | -9.4 (5.42) | -8.1 (5.49)
  Week 8: number analyzed (Participants) | 94 | 96
  Week 8 | -12.0 (5.98) | -10.3 (5.55)
  Week 12: number analyzed (Participants) | 92 | 93
  Week 12 | -14.2 (5.88) | -12.4 (6.02)

6. Secondary Outcome: Change From Baseline in Atopic Dermatitis Control Tool (ADCT) Score at Weeks 2, 4, 8 and 12: Main Study
Description: ADCT score is used to measure the participants perceived AD control. It consists of 6 questions (overall severity of symptoms, days with intense episodes of itching, intensity of bother, problem with sleep, impact on daily activities, and impact on mood or emotions) which are evaluated over the past week on scale from 0 to 4. Scores from all 6 questions are added up to provide ADCT score, ranging from 0 to 24, where higher scores indicate lower AD control.
Time Frame: Baseline (prior to dosing on Day 1), Weeks 2, 4, 8 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Main Study: Abrocitinib 200 mg | Main Study: Abrocitinib 100 mg
Number analyzed (Participants) | 100 | 100
Units on a scale
  Week 2: number analyzed (Participants) | 97 | 98
  Week 2 | -5.2 (4.06) | -4.4 (4.57)
  Week 4: number analyzed (Participants) | 96 | 96
  Week 4 | -8.1 (4.90) | -7.4 (4.64)
  Week 8: number analyzed (Participants) | 94 | 96
  Week 8 | -10.7 (4.80) | -9.4 (5.21)
  Week 12: number analyzed (Participants) | 91 | 93
  Week 12 | -12.8 (5.33) | -11.5 (5.64)

7. Secondary Outcome: Percentage of Participants With Bone Safety Findings in Knee Magnetic Resonance Imaging (MRI) at 1 Year After Randomization: Substudy
Description: MRI imaging session was performed when participant was in supine position in the confined space of the MRI scanner for approximately 30 mins. The assessments included evaluation of epiphyseal plate closure and mineralization of cartilage at the growth centers.
Time Frame: Up to 1 year from randomization on Day 1 of main study
Population: Substudy analysis set included all participants who entered the substudy and who took at least 1 dose of study intervention during the substudy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy: Abrocitinib 100 mg | Substudy: Abrocitinib 200 mg
Number analyzed (Participants) | 19 | 16
Percentage of participants | 0 [0.0 to 17.6] | 0 [0.0 to 20.6]

ADVERSE EVENTS:
Time Frame: Main Study: From Day 1 of dosing up to 4 weeks post last dose (last dose at Week 12, maximum follow-up till Week 16); Sub Study: From Day 1 of dosing (in main study) up to 4 weeks post last dose (last dose at Year 1, maximum follow-up till Year 1.08)
Description: Same event may appear as both AE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. MedDRA version 26.0 was used for main study and 27.0 was used for substudy. Safety analysis set for Main study and substudy analysis set for substudy was evaluated.
Groups:
- Main Study: Abrocitinib 200 mg QD: Participants received abrocitinib 200 mg, orally QD for 12 weeks.
Arm/Group | Main Study: Abrocitinib 200 mg QD | Main Study: Abrocitinib 100 mg QD | Substudy: Abrocitinib 100 mg | Substudy: Abrocitinib 200 mg
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/101 | 0/19 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/99 | 1/101 | 0/19 | 0/16
Other Adverse Events (participants affected / at risk) | 22/99 | 20/101 | 8/19 | 5/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Abrocitinib 200 mg QD (N=99) | Main Study: Abrocitinib 100 mg QD (N=101) | Substudy: Abrocitinib 100 mg (N=19) | Substudy: Abrocitinib 200 mg (N=16)
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Main Study: Abrocitinib 200 mg QD (N=99) | Main Study: Abrocitinib 100 mg QD (N=101) | Substudy: Abrocitinib 100 mg (N=19) | Substudy: Abrocitinib 200 mg (N=16)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 5 | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0/0 | 0/0
Pyrexia (General disorders) | 1 | 3 | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Eczema herpeticum (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Joint tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pyoderma (Infections and infestations) | 0 | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 1

LIMITATIONS AND CAVEATS:
One participant was randomized to abrocitinib 200 mg arm but received abrocitinib 100 mg, hence for safety analysis set of main study that participant was included in 100 mg arm and for full analysis set that participant was included in 200 mg arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT05375929/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT05375929/SAP_001.pdf